CLINICAL TRIAL: NCT01878253
Title: Multicenter Trial of the Sidus Stem-Free Shoulder Arthroplasty System
Brief Title: Sidus Stem-Free Shoulder IDE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIU2012-12E; G130026 (Other: FDA)
Record Dates: First submitted 2013-05-23; First posted 2013-06-14 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis; Posttraumatic Arthrosis; Rheumatoid Arthritis
Keywords: Total Shoulder Arthoplasty
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Investigational (Experimental): This arm will include all subjects who are implanted with the investigational Sidus Stem-Free Total Shoulder Arthroplasty System.
  Interventions: Device: Sidus Stem-Free Total Shoulder Arthroplasty System

INTERVENTIONS:
Device: Sidus Stem-Free Total Shoulder Arthroplasty System

SUMMARY:
The purpose of this study is to determine if Sidus stem-free shoulder system is safe and effective when used in total shoulder replacement.

DETAILED DESCRIPTION:
The primary objectives of this study are to evaluate the safety and efficacy (defined as follows) of the Sidus Stem-Free Shoulder System in unilateral primary total shoulder arthroplasty.

Safety: Will be evaluated by monitoring the frequency and incidence of device related adverse events or unanticipated adverse device effects (UADEs) in investigational subjects as well as analyzing survivorship using revision or intended revision as an endpoint.

Efficacy: Will be determined by comparing the overall pain and functional performance, survivorship and radiographic success of investigational subjects with those subjects who received the control devices.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 22 years of age or older.
* Patient is skeletally mature.
* Patient must have signed the IRB/EC approved informed consent.
* Patient is a candidate for a total shoulder arthroplasty (replacement of humeral head and glenoid).
* Patient has a diagnosis of primary osteoarthritis of the shoulder of grade III or higher.
* Patient has experienced symptoms of shoulder pain and/or loss of function for at least 6 months and has a maximum ASES score of 40.
* Patient has no findings to indicate an etiology of acute trauma, infection, avascular necrosis or inflammatory arthropathy of the operative shoulder.
* Patient has undergone no previous reconstructive shoulder surgery. Acceptable previous shoulder surgeries include arthroscopy, soft tissue repair, or pinning/screw fixation due to a historic fracture.
* Patient is willing and able to comply with the required post-operative therapy as defined in the protocol.
* Patient is willing and able to comply with the required follow-up schedule as defined in the protocol.

Exclusion Criteria:

* Patient is a prisoner.
* Patient is a known current alcohol or drug abuser.
* Patient has a psychiatric illness or cognitive deficit that precluded informed consent.
* Patient has a chronic renal impairment or failure.
* Patient sensitivity to implant materials.
* Patient has a vascular insufficiency due to large or small vessel disease which could inhibit postoperative healing.
* Patient is currently receiving or has received within the last 3 months chronic systemic or inhaled steroids. This exclusion does not apply to those patients with occasional inhaler use due to seasonal allergies.
* Local rash or skin infection around the intended operative site.
* Patients with ongoing Worker's Compensation or third party liability claims related to the operative shoulder.
* Pre-existing contra-lateral shoulder replacement less than 6 months ago.
* Patient who will require a contra-lateral shoulder replacement less than 6 months from the current planned shoulder replacement.
* Patient has evidence of major joint trauma, infection, avascular necrosis, cuff tear arthropathy, chronic dislocation, massive rotator cuff tear, inflammatory arthropathy, or previous shoulder surgery (other than arthroscopy, soft tissue repair, or pinning/screw fixation due to historic fracture).
* Patient has significant muscle paralysis.
* Patient has Charcot arthropathy.
* Patient has metaphyseal bony defects at the bone/implant interface which could inhibit prosthesis fixation.
* Patient has a preoperative computed tomography scans or other radiographic images of the shoulder that showed insufficient glenoid or humeral bone stock to allow for implantation of the prosthesis.
* Insufficient bone stock exists in the presence of metabolic bone disease (i.e. osteoporosis or severe osteopenia), cancer and radiation.
* Patient with severe glenoid deficiency.
* Prior fracture of the operative shoulder with the presence of malunion or non-union.
* Prior tuberosity fracture with the presence of malunion or non-union.
* Patient has an active joint or systemic infection.
* Patient has a life expectancy of less than two years.
* Patient with unacceptably high operative risk.
* Patient unwilling to sign protocol required informed consent.
* Patient is unwilling to complete the protocol required radiographic imaging.
* Patient is unwilling to complete the protocol required follow-up of two years.
* Patient is known to be pregnant.
* Intraoperative findings which indicate insufficient bone stock or local deformities which could inhibit prosthesis fixation. Final assessment of bone quality will be completed intraoperatively upon resection of the humeral head and prior to insertion of the anchor as described in the surgical technique. If there is any doubt regarding bone quality affecting the stable fixation of the anchor, the surgeon must use a stemmed prosthesis.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-07; Primary Completion 2018-05 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (8):
  - Stanford University, Redwood City, California
  - University of California San Francisco - Orthopaedics Institute, San Francisco, California
  - St. Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Norton Orthopaedic & Sports Medicine, Louisville, Kentucky
  - MedStar Health, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Rothman Institute, Philadelphia, Pennsylvania
- Canada (3):
  - University of Calgary Sports Medicine Clinic, Calgary, Alberta
  - Kingston General Hospital, Kingston, Ontario
  - St. Joseph's Health Care London - Hand and Upper Limb Centre, London, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Sidus Stem-Free Shoulder System: This arm will include all subjects who are implanted with the investigational Sidus Stem-Free Total Shoulder Arthroplasty System.
  Sidus Stem-Free Total Shoulder Arthroplasty System
Period: Overall Study
Arm/Group | Sidus Stem-Free Shoulder System
Started | 95
Pre-Operative | 95
6 Weeks | 95
6 Months | 90
1 Year | 88
2 Year | 86
Completed | 86
Not Completed | 9
Not completed — Death | 1
Not completed — SIdus System Removal | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Completed Study w/o Follow-up Data | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sidus Stem-Free Shoulder System
Number analyzed (Participants) | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 55
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 87
  African American | 4
  Asian | 1
  Hispanic or Latino | 1
  Patient Unwilling to Answer | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.8 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Pain and Function as Measured by the American Society of Shoulder and Elbow Surgeons Questionnaire
Description: Pain and function as measured by the American Society of Shoulder and Elbow Surgeons questionnaire. ASES consists of 3 subcomponent scores including pain, instability and activities of daily living. The pain score can be 0 to 10 with 0 being no pain and 10 being the worst pain imaginable. The instability score can be 0 to 10 with 0 being no instability and 10 being the worst instability imaginable. The activities of daily living consists of 10 questions with ordinal responses of 0, 1, 2, and 3. 3 involves no limitation and 0 is unable to do. The 3 subcomponents combine to make the overall ASES score which can range from 0 to 100 with 0 being the worst possible score and 100 being the best.
Time Frame: Two years
Population: All participants received the implant as treatment. ASES Functional Score Summary and Pain Scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sidus Stem-Free Shoulder System: This arm will include all subjects who are implanted with the investigational Sidus Stem-Free Total Shoulder Arthroplasty System.
  Sidus Stem-Free Total Shoulder Arthroplasty System. ASES Functional and Pain Summary scores
Arm/Group | Sidus Stem-Free Shoulder System
Number analyzed (Participants) | 86
score on a scale
  ASES Functional Score | 89.4 (13.3)
  ASES Pain Score | 0.7 (1.5)

2. Primary Outcome: Absence of Radiographic Evidence of Failure or Pending Failure Based on Radiographic Assessment
Description: absence of radiographic evidence of pending failure of the humeral components, assessed at 2 years which may include the following:
  * implant fracture
  * progressive implant migration or subsidence ≥ 5 mm
Time Frame: Two years
Population: Participants who had received the implant. 85 subjects had radiographic images available at the 2 year time point.. Radiographies were assessed at 2 years for implant fracture, failure of humeral components and progressive implant migration or subsidence greater or equal to 5 mm.
Measure: Count of Participants; unit: Participants
Groups:
- Sidus Stem-Free Shoulder System: Absence of radiographic evidence of pending failure of the humeral components, assessed at 2 years which may include the following:
  * implant fracture
  * progressive implant migration or subsidence ≥ 5 mm
Arm/Group | Sidus Stem-Free Shoulder System
Number analyzed (Participants) | 85
Participants
  Subjects with Evidence of Radiographic Failure | 2
  Subjects with Radiographic Success | 83

3. Primary Outcome: The Number of Device Related Serious Adverse Events.
Description: This outcome will measure the frequency of device related serious adverse events.
Time Frame: Two years
Population: This outcome will measure the frequency of device related serious adverse events. At the two year endpoint of the study there were a total of 86 participants with available data.
Measure: Number; unit: Device Related Serious Adverse Events
Groups:
- Investigational: Frequency of device related serious adverse events
Arm/Group | Investigational
Number analyzed (Participants) | 86
Device Related Serious Adverse Events | 0

4. Primary Outcome: Survivorship
Description: The Kaplan-Meier method was used for this study. This outcome measures survivorship of the implanted devices from the date of implantation to the date of revision or intended revision up to 2 years post-operative (whichever came first).
Time Frame: Up to Two years
Population: At the two year study endpoint there were 86 subjects that had data available at the two year time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Sidus Stem-Free Shoulder System
Number analyzed (Participants) | 86
Participants
  Subject devices that survived | 83
  Subject devices revised | 3

5. Secondary Outcome: ASES Functional and Pain Scores at Intervals Other Than 2 Years as Measured by the American Society of Shoulder and Elbow Surgeons Questionnaire
Description: as for outcome 1
Time Frame: 6 weeks, 6 months, and 1 year
Population: ASES Functional Score Summary and Pain Scores. 95 Participants had ASES data at 6 weeks, 90 at 6 months and 88 at 1 year. At 6 weeks 1 subject was missing data required to calculate the ASES functional score, had pain score data present.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sidus Stem-Free Shoulder System: This arm will include all subjects who are implanted with the investigational Sidus Stem-Free Total Shoulder Arthroplasty System.
  Sidus Stem-Free Total Shoulder Arthroplasty System. ASES Functional Summary scores
Arm/Group | Sidus Stem-Free Shoulder System
Number analyzed (Participants) | 95
score on a scale
  ASES Functional Score 6 Weeks: number analyzed (Participants) | 94
  ASES Functional Score 6 Weeks | 59.8 (18.2)
  ASES Functional Score 6 Months: number analyzed (Participants) | 90
  ASES Functional Score 6 Months | 80.3 (20.1)
  ASES Functional Score 1 Year: number analyzed (Participants) | 88
  ASES Functional Score 1 Year | 88.1 (14.5)
  ASES Pain Score 6 weeks | 2 (2.4)
  ASES Pain Score 6 months: number analyzed (Participants) | 90
  ASES Pain Score 6 months | 1.3 (2.2)
  ASES Pain Score 1 year: number analyzed (Participants) | 88
  ASES Pain Score 1 year | 0.7 (1.5)

6. Secondary Outcome: SF-12 Mental Health and Physical Composite Scores as Measured by the SF-12 Scoring Questionnaire.
Description: SF-12 Mental Health and Physical Composite Scores. SF-12 is a validated health survey that uses 12 questions to measure functional health and well being from the patient's point of view. The SF-12 is calculated on a scale of 0 to 100, where a 0 is the worst level of health and 100 is the best level of health. The scores are then normalized with a mean score of 50 and a standard deviation of 10, so that scores greater than 50 represent a health level better than average, and scores less than 50 represent a level lower than average.
Time Frame: Pre-Op, 6 weeks, 6 months, 1 year and 2 years
Population: SF-12 Mental Health and Physical Composite Scores. 95 subjects had data Pre-operatively, 94 at 6 weeks, 90 at 6 months, 88 at 1 year and 86 at 2 years. One subject at the 6 weeks interval had completed the physical portion of the SF-12 but did not complete all requirements to calculate the SF-12 Mental Score.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sidus Stem-Free Shoulder System: This arm will include all subjects who are implanted with the investigational Sidus Stem-Free Total Shoulder Arthroplasty System.
  Sidus Stem-Free Total Shoulder Arthroplasty System SF-12 Mental Health and Physical Composite Scores
Arm/Group | Sidus Stem-Free Shoulder System
Number analyzed (Participants) | 95
score on a scale
  SF-12 Mental Health Scores Pre-Op | 50 (13.5)
  SF-12 Mental Health Scores 6 Weeks: number analyzed (Participants) | 93
  SF-12 Mental Health Scores 6 Weeks | 55.1 (10.5)
  SF-12 Mental Health Scores 6 Months: number analyzed (Participants) | 90
  SF-12 Mental Health Scores 6 Months | 55.5 (8.4)
  SF-12 Mental Health Scores 1 Year: number analyzed (Participants) | 88
  SF-12 Mental Health Scores 1 Year | 54.3 (9.1)
  SF-12 Mental Health Scores 2 Year: number analyzed (Participants) | 86
  SF-12 Mental Health Scores 2 Year | 54.3 (8.3)
  SF-12 Physical Composite Scores Pre-Op | 32.7 (6.9)
  SF-12 Physical Composite Scores 6 weeks: number analyzed (Participants) | 94
  SF-12 Physical Composite Scores 6 weeks | 36.5 (8.3)
  SF-12 Physical Composite Scores 6 months: number analyzed (Participants) | 90
  SF-12 Physical Composite Scores 6 months | 44.2 (10.6)
  SF-12 Physical Composite Scores 1 year: number analyzed (Participants) | 88
  SF-12 Physical Composite Scores 1 year | 46.2 (10.3)
  SF-12 Physical Composite Scores 2 year: number analyzed (Participants) | 86
  SF-12 Physical Composite Scores 2 year | 47.6 (8.7)

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events from the date each subject was implanted until the date of study closure or date of revision (if applicable).
Description: If a subject experienced more than 1 of a given AE, the subjects are counted only once for that AE. If a subject experienced more than one AE in a system organ class (SOC), the subject is counted only once in that SOC.
Arm/Group | Sidus Stem-Free Shoulder System
All-Cause Mortality (participants affected / at risk) | 1/95
Serious Adverse Events (participants affected / at risk) | 0/95
Other Adverse Events (participants affected / at risk) | 28/95
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sidus Stem-Free Shoulder System (N=95)
Dermatological (Skin and subcutaneous tissue disorders) | 1 (1) — Chronic Urticarial
Other General Non-Shoulder Complication (Musculoskeletal and connective tissue disorders) | 5 (11) — Abnormal Radiographic Findings
Fracture of Proximal Humerus (Musculoskeletal and connective tissue disorders) | 1 (1) — Fracture of Proximal Humerus During Surgery
Glenoid Implant Loosening (Musculoskeletal and connective tissue disorders) | 3 (3) — Post-operative Glenoid Implant Loosening
Other Shoulder Related Complication (Musculoskeletal and connective tissue disorders) | 21 (29) — Other non-specified shoulder complication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator must provide the Sponsor at least 30 days to review publications for legal and regulatory compliance and will include in publications a statement that the study was supported by the Sponsor. Sponsor confidential information will not be submitted for publication without Sponsor consent. Sponsor may request delay of publication for 60 days to allow for patent application filing.

DOCUMENTS (1):
  • Study Protocol (2013-07-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT01878253/Prot_000.pdf